# Impact of Consumption of Beta-glucans on the Intestinal Microbiota and Glucose and Lipid Metabolism

ClinicalTrials.gov registration number: NCT02041104

### Study performed by:

Ana Velikonja<sup>a</sup>, Luka Lipoglavšek<sup>b</sup>, Rok Orel<sup>c</sup>, Gorazd Avguštin<sup>b\*</sup>

Study was sponsored by the company Mlinotest d.d., Ajdovščina, Slovenia and by the research programme P4-0097 of the Slovenian Research Agency

<sup>&</sup>lt;sup>a</sup> Mlinotest d.d., Tovarniška cesta 14, SI-5270 Ajdovščina, Slovenia

<sup>&</sup>lt;sup>b</sup> University of Ljubljana, Biotechnical Faculty, Department of Animal Science, Groblje 3, SI-1230 Domžale, Slovenia

<sup>&</sup>lt;sup>c</sup> University Medical Centre Ljubljana, University Children`s Hospital, Department of Gastroenterology, Hepatology and Nutrition, Bohoričeva 20, SI-1000 Ljubljana, Slovenia

#### STUDY PROTOCOL

»Impact of Consumption of Beta-glucans on the Intestinal Microbiota and Glucose and Lipid Metabolism«

#### Introduction

Metabolic syndrome (MS) is a complex lifestyle disease manifesting metabolic disorders such as abdominal obesity, dyslipidemia, hyperglycemia and hypertension. There are many studies reporting how gut microbiota correlates with metabolic disorders or contributes to the development of obesity trough increased energy harvest. An increasing interest in finding the diet that could regulate the composition of gut microbiota and consequently improve the individual conditions related to some of the metabolic disorders, exists. The aim of our study will be to investigate, whether consumption of barley beta glucans can positively modulate the composition of gut microbiota and metabolic parameters related to MS. Barley beta glucans are polysaccharides found in kernel endosperm and improve both lipid and glucose metabolism. The effects of barley beta glucans on gut microbiota composition are still poorly investigated in human clinical trials.

We will perform a double-blind, placebo controlled, randomized clinical trial with volunteers diagnosed with MS. The exact study protocol and procedure will be explained to the participants, who will meet inclusion criteria. After assignment of participation agreement, participant will be randomized and allocated to test or placebo group. Before and after the dietary intervention, anthropometric measurements, blood analysis, including oral glucose tolerance testing (OGTT), and fecal sampling will be performed. Participants will daily complete food frequency questionnaire and detailed 72-hour dietary recall. During intervention participants will daily consumed test bread with added 6g beta glucans or bread without added beta-glucans.

The study was approved by the Republic of Slovenia National Medical Ethics Committee (112/08/13).

### **Study protocol**

## A) Participants information and inclusion criteria

| Name |
|-------------------------------------------------------|
| Surname |
| Age |
| Body height & body weight (cm, kg) |
| Diabetes type 2 |
| Kidney disfunction |
| Thyroid disfunction |
| Treatment for hypercholesterolemia (not hypertension) |
| Total cholesterol (mmol /l) |
| Body Mass Index (BMI) |

# B) Before and after intervention: Blood test Analysis and Anthropometric measurements

### 1. Lipid profile, Anthropometric measurements

| Parameter | Before dietary intervention | After dietary intervention |
|---|---|---|
| Total cholesterol (mmol/l) | | |
| LDL-cholesterol (mmol/l) | | |
| HDL-cholesterol (mmol/l) | | |
| Triglycerides (mmol/l) | | |
| Blood pressure (mmHg) | | 1 |
| Body weight (kg) | | |
| Body waist (cm) | | |

## 2. Oral glucose tolerance test (OGTT)

| Sampling | Before dietary intervention | | After dietary intervention | |
|---|---|---|---|---|
| time after | Glucose level | Insulin level | Glucose level | Insulin level |
| glucose | (mmol/l) | (μU/ml) | (mmol/l) | (µU/ml) |
| consumption | | | | |
| (min) | | | | |
| 0 | | | | |
| 30 | | | | |
| 60 | | | | |
| 120 | | | | |

### 3. Gut microbiota analysis and short chain fatty acids measurements

Faecal samples will be obtained before and after dietary intervention.

Analysis of gut microbiota composition will be performed followed DNA extraction, with several methodologies; Denaturing Gradient Gel Electrophoresis (DGGE), qPCR, new generation sequencing (illumine Miseq platform).

### **Short-chain fatty acids determination**

| Short-chain fatty acid | Before dietary intervention (g/kg) | After dietary intervention (g/kg) |
|---|---|---|
| Butyric acid | | |
| Acetic acid | | |
| Propionic acid | | |

# 4. 72-hour dietary recall

Dietary recall will be performed three times before and during dietary intervention to obtain average nutrient intake:

| Average nutrition intake | Before dietary | Between dietary |
|--------------------------|----------------|-----------------|
| per 100 g | intervention | intervention |
| Energy (kcal) | | |
| Protein (g) | | |
| Fat (g) | | |
| Total carbohydrates (g) | | |
| Total dietary fibre (g) | | |
| Water (g) | | |